CLINICAL TRIAL: NCT02443831
Title: Immunotherapy with CD19+CD22 CAR Redirected T-cells for High Risk/relapsed Paediatric CD19+ and CD22+ Acute Lymphoblastic Leukaemia
Brief Title: CARPALL: Immunotherapy with CD19+CD22 CAR T-cells for CD19+ and CD22+ Acute Lymphoblastic Leukaemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL 14/0529
Record Dates: First submitted 2015-04-29; First posted 2015-05-14 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: high risk relapsed CD19+ and CD22+ acute lymphoblastic leukaemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Leukapheresis; Whole-Body Irradiation; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19+CD22 CAR T-cells (Experimental): Patients meeting the eligibility criteria will have leukapheresis to isolate the blood immune cells used to manufacture the CD19+CD22CAR T-cells. Patients will receive lymphodepletion with low dose total body irradiation, fludarabine and cyclophosphamide prior to infusion of the CD19+CD22CAR T-cells.
  Interventions: Procedure: Leukapheresis; Radiation: Total Body Irradiation (TBI); Drug: Lymphodepletion with Fludarabine; Drug: Lymphodepletion with Cyclophosphamide; Biological: CD19+CD22 CAR T-cells

INTERVENTIONS:
Procedure: Leukapheresis — Patients will undergo an unstimulated leukapheresis to isolate the required immune cells to produce the CD19+CD22 CAR T-cells
Radiation: Total Body Irradiation (TBI) — Participants will receive total body irradiation delivered as a single fraction (2Gy) on day -7 prior to CD19+CD22CAR T-cell infusion.
Drug: Lymphodepletion with Fludarabine — Patients will receive lymphodepleting chemotherapy with iv fludarabine 30 mg/m2 on days -6 to -3 prior to CD19+CD22CAR T-cell infusion.
Drug: Lymphodepletion with Cyclophosphamide — Patients will receive lymphodepleting chemotherapy with iv cyclophosphamide 0.5 g/m2 on days -6 to -5 prior to CD19+CD22CAR T-cell infusion.
Biological: CD19+CD22 CAR T-cells — Dose level 1: 2 doses of 4 x 10^5 CD19+CD22 CAR T-cells/kg Dose level 2: 2 doses of 1 x 10^6 CD19+CD22 CAR T-cells/kg given as a split dose as an intravenous injection through a Hickman line or PICC line (peripherally inserted central catheter) on day 0 and day 14.

SUMMARY:
This study aims to evaluate the safety, efficacy and duration of response of CD19+CD22 Chimeric Antigen Receptor (CAR) redirected autologous T-cells in children with high risk, relapsed CD19+ and CD22+ acute lymphoblastic leukaemia

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product named CD19+CD22 Chimeric Antigen Receptor (CAR) T-cells (CD19+CD22 CAR T-cells) in children and young adults (age <24 years) with high risk, relapsed CD19+ and CD22+ acute lymphoblastic leukaemia. Following informed consent and registration to the trial, patients will undergo an unstimulated leukapheresis for the generation of the CD19+CD22 CAR T-cells. Patients will receive the CD19+CD22CAR T-cells following lymphodepleting chemotherapy and total body irradiation. The study will evaluate the safety, efficacy and duration of response of the CD19+CD22 CAR T-cells in children with high risk relapsed CD19+ and CD22+ acute lymphoblastic leukaemia.

ELIGIBILITY:
Inclusion Criteria:

1. Children and young adults (age 24 years or younger) with high risk/relapsed CD19+ and CD22+ acute lymphoblastic leukaemia with:

   1. Resistant disease (>5% blasts) at end of ALLTogether-1 protocol or equivalent induction
   2. ALL with persisting high level MRD at 2nd time point of frontline national protocol (currently MRD >10-4 at week 9 ALLTogether-1 Protocol or equivalent).
   3. High risk infant ALL (age < 6 months at diagnosis with MLL gene rearrangement and either presenting white cell count > 300 x 10^9/L or poor steroid early response (i.e. circulating blast count >1x10^9/L following 7 day steroid pre-phase of induction as per national guidelines or equivalent)
   4. Any patient with t(17,19) TCF3-HLF rearrangement
   5. High risk 1st relapse (defined as very early (relapse within 18 months of diagnosis) and early relapses (any patient relapsing on therapy or within 6 months of completing treatment) and any relapse with high risk genetics, namely (KMT2A (MLL) rearrangements, low hypodiploidy/near haploidy, t(17;19)(q22;p13)/TCF3-HLF, iAMP21 and t(1;19)(q21;p13)/TCF3- PBX1, t(9;22)(34.1 q11.2)/BCR-ABL1
   6. Any on therapy relapse in patients age 16-24
   7. Any relapse of infant ALL
   8. ALL post ≥ 2nd relapse
   9. Any refractory relapse of ALL (defined as > 1% blasts by flow cytometry after a at least 1 cycle of standard chemotherapy)
   10. ALL with MRD >10-4 prior to planned stem cell transplant
   11. Any relapse of ALL eligible for stem cell transplant but no available HLA matched donor or other contraindication to transplant
   12. Any relapse of ALL after stem cell transplant as long as planned time of CD19+CD22CAR T cell infusion is > 4 months post-transplant
   13. Early (defined as < 6 months post-infusion) loss of B cell aplasia or any CD19+CD22+ relapse following CD19CAR T cell therapy with Tisagenlecleucel

   Note patients with isolated CNS relapse meeting one or more of the criteria above are eligible for the study
2. Agreement to have a pregnancy test, use adequate contraception (if applicable)
3. Written informed consent

Exclusion Criteria:

Exclusion Criteria for registration:

1. Active Hepatitis B, C or HIV infection
2. Oxygen saturation ≤ 90% on air
3. Bilirubin > 3 x upper limit of normal
4. Creatinine > 3 x upper limit of normal
5. Women who are pregnant or breastfeeding
6. Stem Cell Transplant patients only: active significant (overall Grade ≥ II, Seattle criteria) acute GVHD or moderate/ severe chronic GVHD (NIH consensus criteria) requiring systemic steroids.
7. Inability to tolerate leucapheresis
8. Karnofsky (age ≥ 10 years) or Lansky (age < 10) score ≤ 50%
9. Pre-existing significant neurological disorder (other than CNS involvement of underlying haematological malignancy)
10. CD19 negative or CD22 negative disease

Exclusion criteria for CD19+CD22CAR T-cell infusion:

1. Severe intercurrent infection at the time of scheduled CD19+CD22 CAR T-cell infusion
2. Requirement for supplementary oxygen or active pulmonary infiltrates at the time of scheduled CD19+CD22 CAR T-cell infusion
3. Allogeneic transplant recipients with active significant acute GVHD overall grade ≥II or moderate/severe chronic GVHD requiring systemic steroids at the time of scheduled CD19+CD22 CAR T-cell infusion. Note: Such patients will be excluded until the patient is GVHD free and off steroids

In addition, for CAR T infusion on D14: absence of CRS>Gr2 or ICANS>Gr2 after D0 CAR T infusion.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) following CD19+CD22 CAR T-cell infusion | 28 days
  The incidence of dose limiting toxicity (DLT) occurring within 28 days of CD19+CD22CAR T-cell infusion.
Molecular remission | 28 days
  Efficacy will be assessed by determining Minimal Residual Disease in the bone marrow aspirate using immunoglobulin heavy chain (IgH) quantitative polymerase chain reaction (qPCR) and/or Next Generation Sequencing in all patients. The proportion of patients achieving molecular remission at 28 days post CD19+CD22CAR T-cell infusion will be determined.

SECONDARY OUTCOMES:
Feasibility of Generation of CD19+CD22 CAR T-cells | Day 28
  Evaluated by the number of therapeutic products generated.
Molecular Remission | 3 months
  Efficacy will be assessed by determining Minimal Residual Disease in the bone marrow aspirate using immunoglobulin heavy chain (IgH) quantitative polymerase chain reaction (qPCR) and/or Next Generation Sequencing in all patients. The proportion of patients achieving molecular remission at 3 months post CD19+CD22CAR T-cell infusion will be determined.
Long-Term Molecular Remission | 2 years
  Number of patients in molecular remission without further therapy at 1 and 2 years
Duration of Response | 15 years
  Duration of response is measured from the time of achieving molecular remission or flow MRD negativity until the disease relapse or death, whichever occurs first.
Safety and Tolerability of the CAR T-cells | 15 years
  Incidence of adverse events and reactions (toxicity) to the CAR T-cells.
Incidence of B Aplasia | 2 years
  Incidence of B aplasia
Incidence of Hypogammaglobulinaemia | 2 years
  Incidence of hypogammaglobulinaemia
Frequency of Circulating CD19+CD22 CAR T-cells | 2 years
  Persistence and frequency of circulating CD19+CD22CAR T-cells in the peripheral blood by flow cytometry and qPCR analyses.
Relapse rate | 2 years
  Relapse rate
Overall Survival (OS) | 2 years
  Overall Survival (OS) at 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Persis Amrolia, Study Chair — UCL Institute of Child Health
Locations (3):
- United Kingdom (3):
  - Great Ormond Street Hospital, London
  - University College Hospital, London
  - Manchester Royal Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghorashian S, Lucchini G, Richardson R, Nguyen K, Terris C, Guvenel A, Oporto-Espuelas M, Yeung J, Pinner D, Chu J, Williams L, Ko KY, Walding C, Watts K, Inglott S, Thomas R, Connor C, Adams S, Gravett E, Gilmour K, Lal A, Kunaseelan S, Popova B, Lopes A, Ngai Y, Hackshaw A, Kokalaki E, Carulla MB, Mullanfiroze K, Lazareva A, Pavasovic V, Rao A, Bartram J, Vora A, Chiesa R, Silva J, Rao K, Bonney D, Wynn R, Pule M, Hough R, Amrolia PJ. CD19/CD22 targeting with cotransduced CAR T cells to prevent antigen-negative relapse after CAR T-cell therapy for B-cell ALL. Blood. 2024 Jan 11;143(2):118-123. doi: 10.1182/blood.2023020621. PMID 37647647
- [Derived] Kokalaki E, Ma B, Ferrari M, Grothier T, Hazelton W, Manzoor S, Costu E, Taylor J, Bulek A, Srivastava S, Gannon I, Jha R, Gealy R, Stanczuk L, Rizou T, Robson M, El-Kholy M, Baldan V, Righi M, Sillibourne J, Thomas S, Onuoha S, Cordoba S, Pule M. Dual targeting of CD19 and CD22 against B-ALL using a novel high-sensitivity aCD22 CAR. Mol Ther. 2023 Jul 5;31(7):2089-2104. doi: 10.1016/j.ymthe.2023.03.020. Epub 2023 Mar 21. PMID 36945773
- [Derived] Ghorashian S, Kramer AM, Onuoha S, Wright G, Bartram J, Richardson R, Albon SJ, Casanovas-Company J, Castro F, Popova B, Villanueva K, Yeung J, Vetharoy W, Guvenel A, Wawrzyniecka PA, Mekkaoui L, Cheung GW, Pinner D, Chu J, Lucchini G, Silva J, Ciocarlie O, Lazareva A, Inglott S, Gilmour KC, Ahsan G, Ferrari M, Manzoor S, Champion K, Brooks T, Lopes A, Hackshaw A, Farzaneh F, Chiesa R, Rao K, Bonney D, Samarasinghe S, Goulden N, Vora A, Veys P, Hough R, Wynn R, Pule MA, Amrolia PJ. Enhanced CAR T cell expansion and prolonged persistence in pediatric patients with ALL treated with a low-affinity CD19 CAR. Nat Med. 2019 Sep;25(9):1408-1414. doi: 10.1038/s41591-019-0549-5. Epub 2019 Sep 2. PMID 31477906